CLINICAL TRIAL: NCT05072145
Title: Evaluating the Role of Tele-Emergency Care in Health Care Costs and Long-Term Outcomes for Rural Medicare Beneficiaries With Sepsis
Brief Title: Evaluating Tele-Emergency Care in Costs and Outcomes for Rural Sepsis Patients
Acronym: TELE-Cost
Status: Completed | Type: Observational
Sponsor: Nicholas M Mohr (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Nicholas M Mohr, Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202011064
Record Dates: First submitted 2021-09-08; First posted 2021-10-08 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Sepsis
Keywords: Telemedicine
MeSH Terms: conditions — Sepsis | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-tele-ED hospital: Patients receiving care in an ED that does not provide any tele-ED service
- Tele-ED hospital: Patients receiving care in an ED that uses tele-ED services, but patient care did NOT utilize this service
- Tele-ED used: Patient care was provided through tele-ED services
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — Receiving care in a tele-ED hospital
  Groups: Tele-ED used

SUMMARY:
Sepsis is a life-threatening emergency for which provider-to-provider telemedicine has been used to improve quality of care. The objective of this study is to measure the impact of rural tele-emergency consultation on long-term health care costs and outcomes through decreasing organ failure, hospital length-of-stay, and readmissions.

DETAILED DESCRIPTION:
Sepsis is responsible for over 1.7 million hospitalizations at a cost of $26 billion annually, making it the most expensive acute care condition in US hospitals. High-quality early sepsis care has been associated with decreased organ failure, shorter ICU and hospital length-of-stay, and improved survival. Rural sepsis patients are more likely to be transferred to tertiary centers, and they also have higher mortality and health care costs. ED-based telemedicine (tele-ED) consultation between a rural provider and a board-certified emergency physician may deliver the expertise to reduce care delays and improve outcomes while avoiding unnecessary costs.

In 2017, the study team partnered with Avera eCARE, the largest tele-ED provider in North America, to implement a standard telemedicine-based sepsis care pathway. Subsequently, the investigators showed (using patient-level primary data collection across several networks) that tele-ED use was associated with improved adherence with international sepsis guidelines.

In addition to its association with short-term clinical outcomes, however, the study team hypothesize that telemedicine may also decrease costs. The investigators have shown that high-quality sepsis care is associated with decreased readmissions and post-discharge mortality. High quality care may also prevent organ failure, avoid ICU admissions, reduce mechanical ventilation and vasopressor use, decrease ICU and hospital length-of-stay, and decrease post-discharge care-primarily through reducing avoidable organ failure. All of these factors are likely to have a significant effect in terms of reducing healthcare cost.

The objective of the proposed project is to measure the effect of tele-ED consultation at reducing healthcare costs and long-term outcomes in sepsis patients in rural EDs. The following primary hypotheses will be tested:

* Total healthcare expenses and 90-day mortality will be lower in patients treated in a tele-ED hospital, with the effect primarily through reduced hospital length-of-stay and fewer readmissions.
* Total expenses and mortality will be lower in cases where tele-ED is used vs. matched controls in non-tele-ED hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis, according to ICD-10 codes

Exclusion Criteria:

* No infection diagnosed in the ED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age-qualifying Medicare beneficiaries with at least one ED admission for sepsis in a cohort of rural hospitals in the Avera service area between 2017-2019. Hospitals will be stratified as tele-ED capable and a set of 2:1 matched control hospitals in the same regions where tele-ED is not available. Sepsis cases will be identified according to the International (ICD-10), with a discharge diagnosis of [(infection plus organ failure) or explicit sepsis diagnosis], plus an ED diagnosis of infection, as we have done previously.
Sampling Method: Non-Probability Sample
Enrollment: 55772 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Total healthcare expenditures | From hospital admission until 30 days after discharge
  Defined as direct inpatient and outpatient payments to hospitals and physicians, skilled nursing care, home care, durable medical equipment, and ambulance costs from the ED visit until 30 days post-discharge. Drugs are not included.

SECONDARY OUTCOMES:
Number of participants who die within 90 days of hospital admission | From hospital admission until 90 days after admission
  90-day mortality
Hospital length-of-stay | From date of hospitalization through hospital discharge, assessed up to 90 days
  Duration of hospitalization
Number of participants requiring ICU care | From the date of hospital admission through hospital discharge or 90 days, whichever comes first, the number of participants who are treated in an intensive care unit
  Any admission to the ICU
Emergency department costs | From the date of hospital admission through hospital discharge or 90 days, whichever comes first, all emergency department health care expenditures
  Total healthcare expenditures related to emergency department care in current hospitalization
Inpatient care costs | From the date of hospital admission through hospital discharge or 90 days, whichever comes first, all inpatient health care expenditures
  Total healthcare expenditures related to inpatient care in current hospitalizations
Inter-hospital transfer costs | From the date of hospital admission through hospital discharge or 90 days, whichever comes first, all inter-hospital transfer health care expenditures
  Emergency medical services transfer costs and second emergency department costs (if transferred)
Post-discharge costs | From the date of hospital discharge through 30 days after discharge, total health care expenditures health care expenditures
  Total healthcare expenditures
Readmission costs | Between hospital discharge and 30 days after hospital discharge, related to inpatient re-hospitalization
  Total healthcare expenditures during readmission(s) within 30 days after initial hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Mohr, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohr NM, Schuette AR, Ullrich F, Mack LJ, DeJong K, Camargo CA Jr, Zachrison KS, Boggs KM, Skibbe A, Bell A, Pals M, Shane DM, Carter KD, Merchant KA, Ward MM. An economic and health outcome evaluation of telehealth in rural sepsis care: a comparative effectiveness study. J Comp Eff Res. 2022 Jul;11(10):703-716. doi: 10.2217/cer-2022-0019. Epub 2022 May 24. PMID 35608080